CLINICAL TRIAL: NCT04590014
Title: Clinical Efficacy in Relief of Dyspnea by HVNI: Evaluation of New Device Equivalence
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study was not needed from trial standpoint
Sponsor: Vapotherm, Inc. (Industry)
Collaborators: VA Pittsburgh Healthcare System (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: RP-VT2.02020001Sci
Record Dates: First submitted 2020-10-05; First posted 2020-10-19 (Actual); Results first posted 2024-03-20 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-02

CONDITIONS: Dyspnea; Hypercapnia; Respiratory Insufficiency
MeSH Terms: conditions — Dyspnea; Hypercapnia; Respiratory Insufficiency

STUDY DESIGN:
Masking Description: This trial is non-blinded by necessity, as there are distinct differences in size and appearance between the new and current HVNI device designs.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Conventional HVNI First, Then New HVNI Second (Randomized) (Experimental): The purpose of this intervention is to evaluate the efficacy of the conventional HVNI device design (Precision Flow) to provide targeted relief of dyspnea. The purpose of this intervention is to evaluate the efficacy of a new HVNI device design (V2.0) to provide targeted relief of dyspnea.
  Interventions: Device: Conventional Precision Flow; Device: HVNI HVT2.0 Device
- New HVNI First, Then Conventional HVNI Second (Randomized) (Experimental): The purpose of this intervention is to evaluate the efficacy of the conventional HVNI device design (Precision Flow) to provide targeted relief of dyspnea. The purpose of this intervention is to evaluate the efficacy of a new HVNI device design (V2.0) to provide targeted relief of dyspnea.
  Interventions: Device: Conventional Precision Flow; Device: HVNI HVT2.0 Device

INTERVENTIONS:
Device: Conventional Precision Flow — Patients will be placed on HVNI therapy using Vapotherm's conventional HVNI device design (Precision Flow). Patients will receive HVNI therapy through an appropriately-fitted Prosoft dual-pronged nasal cannula. Physiologic and ventilation parameters will be recorded.
  Other Names: Vapotherm Precision Flow
Device: HVNI HVT2.0 Device — Patients will be placed on HVNI therapy using Vapotherm's new HVNI device design (V2.0). Patients will receive HVNI therapy through an appropriately-fitted Prosoft dual-pronged nasal cannula. Physiologic and ventilation parameters will be recorded.
  Other Names: HVNI Device Vapotherm V2.0

SUMMARY:
This study will evaluate the ability of a new High Velocity Nasal Insufflation [HVNI] device design to effect ventilation and related physiological responses relative to the current HVNI device design.

DETAILED DESCRIPTION:
The objective of this study is to evaluate the ability of a new HVNI device to improve ventilation, dyspnea, and related physiological responses relative to the conventional Precision Flow device design, with which there are published clinical outcomes data. It is hypothesized that the new HVNI device design (V2.0) will be comparable at relieving patient dyspnea when compared to the conventional HVNI device design (Precision Flow).

ELIGIBILITY:
Inclusion Criteria:

* Adult inpatients (18 years of age and older)
* Demonstrated severe dyspnea at baseline (Borg Rated Perceived Dyspnea [RPD] (scale 0-10) of 3 or higher)
* Severe baseline hypercarbia/hypercapnia of 55 mmHg or higher as measured by TcPCo2 or arterial or venous blood gas

Exclusion Criteria:

* Patient has unstable cardiovascular condition
* Significant unilateral or bilateral nasal occlusion
* Inability to provide informed consent
* Pregnancy
* Known contraindication to perform steps of the protocol
* Absence of spontaneous respiration or known contraindication to HVNI
* Inability to use HVNI therapy
* Agitation or uncooperativeness
* Determined by the clinician to be sufficiently unstable or unsuitable for this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2022-01-12 (Actual); Primary Completion 2022-07-15 (Actual); Study Completion 2022-07-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles Atwood, Principal Investigator — VA Pittsburgh Healthcare System
Locations (1):
- VA Pittsburgh Healthcare System, Pittsburgh, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Conventional HVNI First New HVNI Second (Randomized): Conventional First, New Second:
  Patients will be placed on HVNI therapy using Vapotherm's conventional HVNI device design (Precision Flow). Patients will receive HVNI therapy through an appropriately-fitted Prosoft dual-pronged nasal cannula. Physiologic and ventilation parameters will be recorded.
  Next, patients will be placed on HVNI therapy using Vapotherm's new HVNI device design (V2.0). Patients will receive HVNI therapy through an appropriately-fitted Prosoft dual-pronged nasal cannula. Physiologic and ventilation parameters will be recorded.
- New HVNI First, Conventional HVNI Second (Randomized): New First, Conventional Second:
  Patients will be placed on HVNI therapy using Vapotherm's new HVNI device design (V2.0). Patients will receive HVNI therapy through an appropriately-fitted Prosoft dual-pronged nasal cannula. Physiologic and ventilation parameters will be recorded.
  Next, patients will be placed on HVNI therapy using Vapotherm's conventional HVNI device design (Precision Flow). Patients will receive HVNI therapy through an appropriately-fitted Prosoft dual-pronged nasal cannula. Physiologic and ventilation parameters will be recorded.
Period: Overall Study
Arm/Group | Conventional HVNI First New HVNI Second (Randomized) | New HVNI First, Conventional HVNI Second (Randomized)
Started | 2 | 3
Completed | 1 | 3
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Conventional HVNI First New HVNI Second (Randomized) | New HVNI First, Conventional HVNI Second (Randomized) | Total
Number analyzed (Participants) | 1 | 3 | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 1 | 3 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 1 | 3 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 1 | 3 | 4
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Patient Vital Signs -- Rated Perceived Dyspnea (RPD)
Description: Patient's subjective assessment of their dyspnea, rated as a modified Borg score on a scale from 0 to 10. Higher scores indicate a worse outcome.
Time Frame: Through study completion, an average of 1.6 hours
Measure: Median (95% Confidence Interval); unit: Units on a scale
Groups:
- Precision Flow: Patients were placed on HVNI therapy using Vapotherm's conventional HVNI device design (Precision Flow)Physiologic and ventilation parameters will be recorded.
- HVT 2.0: Patients were placed on HVNI therapy using Vapotherm's new HVNI device design (HVT 2.0)Physiologic and ventilation parameters will be recorded.
Arm/Group | Precision Flow | HVT 2.0
Number analyzed (Participants) | 4 | 4
Units on a scale
  Baseline | 2.5 [.98 to 4.02] | 3 [.61 to 5.38]
  Therapeutic Characterization once the HVNI settings are having a therapeutic effect. | 2.5 [0.25 to 4.75] | 2 [0.00 to 4.00]

2. Secondary Outcome: Patient Vital Signs - Heart Rate [HR]
Description: Heart rate, measured in beats per minute (bpm)
Time Frame: Through study completion, an average of 1.6 hours
Measure: Median (95% Confidence Interval); unit: bpm
Arm/Group | Precision Flow | HVT 2.0
Number analyzed (Participants) | 4 | 4
bpm
  Baseline | 81 [78.24 to 83.76] | 76.5 [72.32 to 80.68]
  Therapeutic Characterization once the HVNI settings are having a therapeutic effect. | 81.5 [79.98 to 83.02] | 79 [75.47 to 82.53]

3. Secondary Outcome: Patient Vital Signs - Respiratory Rate [RR]
Description: Respiratory rate, measured in breaths per minute (brpm)
Time Frame: Through study completion, an average of 1.6 hours
Measure: Median (95% Confidence Interval); unit: breaths per min
Groups:
- Precision Flow: Patients were placed on HVNI therapy using Vapotherm's conventional HVNI device design (Precision Flow)Physiologic and ventilation parameters will be recorded.cannula. Physiologic and ventilation parameters will be recorded.
Arm/Group | Precision Flow | HVT 2.0
Number analyzed (Participants) | 4 | 4
breaths per min
  Baseline | 19 [11.42 to 26.58] | 17 [12.89 to 21.11]
  Therapeutic Characterization once the HVNI settings are having a therapeutic effect. | 16 [8.94 to 23.06] | 12 [6.49 to 17.51]

4. Secondary Outcome: Patient Vital Signs - Blood Pressure [BP]
Description: Blood pressure (systolic) measured in mmHg
Time Frame: Through study completion, an average of 1.6 hours
Measure: Median (95% Confidence Interval); unit: mmHg
Arm/Group | Precision Flow | HVT 2.0
Number analyzed (Participants) | 4 | 4
mmHg
  Baseline Systolic | 126.5 [108.07 to 144.98] | 125 [90.87 to 159.13]
  Baseline Diastolic | 63 [47.09 to 78.91] | 68.5 [53.61 to 83.29]
  Therapeutic Systolic | 129 [111.70 to 146.30] | 136 [104.46 to 166.54]
  Therapeutic Diastolic | 73.5 [55.15 to 91.85] | 68.5 [57.84 to 79.16]

5. Secondary Outcome: Patient Vital Signs - Arterial Oxygen Saturation [SpO2]
Description: SpO2 measured as percentage of oxygen saturation (%)
Time Frame: Through study completion, an average of 1.6 hours
Measure: Median (95% Confidence Interval); unit: % oxygen
Arm/Group | Precision Flow | HVT 2.0
Number analyzed (Participants) | 4 | 4
% oxygen
  Baseline | 96 [94.00 to 98.00] | 95 [88.85 to 101.15]
  Therapeutic Characterization once the HVNI settings are having a therapeutic effect. | 94.5 [93.58 to 95.42] | 94.5 [90.71 to 98.29]

6. Secondary Outcome: Patient Vital Signs - Transcutaneous CO2 [TcPCO2]
Description: TcPCO2, measured as percentage of CO2 (%)
Time Frame: Through study completion, an average of 1.6 hours
Measure: Median (95% Confidence Interval); unit: % CO2
Arm/Group | Precision Flow | HVT 2.0
Number analyzed (Participants) | 4 | 4
% CO2
  Baseline | 52.1 [30.03 to 74.17] | 54.8 [42.30 to 67.31]
  Therapeutic Characterization once the HVNI settings are having a therapeutic effect. | 49.9 [15.14 to 84.66] | 53.1 [41.36 to 64.84]

ADVERSE EVENTS:
Time Frame: For the duration of the study, from baseline to end of study, which was about 1.65 hours
Description: Any untoward or unfavorable medical occurrence in a participant, including any abnormal sign (for example, abnormal physical exam or laboratory finding), symptom, or disease, temporally associated with the participant's participation in the research, whether or not considered related to the participant's participation in the research.
Arm/Group | Precision Flow | HVT 2.0
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/4
Other Adverse Events (participants affected / at risk) | 0/4 | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-06-11): https://cdn.clinicaltrials.gov/large-docs/14/NCT04590014/Prot_SAP_000.pdf